CLINICAL TRIAL: NCT01497951
Title: A Randomized Controlled Trial: Photodynamic Treatment for the Therapy of Premalignant Mucosal Oral Lesions.
Brief Title: Photodynamic Therapy for Oral Precursor Lesions
Acronym: PDT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dvorak Gabriella, Univ.Ass.DDr., senior staff at department of oral surgery, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010_MuSH
Record Dates: First submitted 2011-12-09; First posted 2011-12-23 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Leukoplakia; Lichen
MeSH Terms: conditions — Leukoplakia | interventions — 5-aminolaevulinic acid-n-pentylester

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aminolaevulinic acid (Experimental)
  Interventions: Other: Aminolaevulinic acid
- Placebo (Placebo Comparator)
  Interventions: Other: Methylcellulose Placebo

INTERVENTIONS:
Other: Aminolaevulinic acid — Photodynamic therapy
  Arms: Aminolaevulinic acid
Other: Methylcellulose Placebo — Methylcellulose
  Arms: Placebo

SUMMARY:
Pre-malignant lesions are difficult to treat. Even after surgical removal they tend to re-appear. Often the lesions are to large and are apparent on many sites, therefore surgical removal is not always possible. The photodynamic therapy uses a special substance, which is absorbed in cells, and thereafter activated by a defined light. The aim of this study is to compare the photodynamic therapy in potentially malignant lesions to a placebo. The investigators assume a significant better result in photodynamic therapy then treatment with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Existing Leukoplakia simplex SIN III (diagnostics by Biopsie)
* Leukoplakia verrucosa without indications of malignant changes (diagnostics by Biopsie)
* Oral Lichen planus SIN III (diagnostics by Biopsie)
* Good mouth hygiene status (tartar, surface)
* Correct seat of the prosthesis and/or the denture
* Located erosions in the oral cavity
* Minimum age:18 years
* Women at the age capable of child-bearing with an appropriate contraception

Exclusion Criteria:

* Malignant changes of the mucous membrane, heavy Dysplasie SIN III, Carcinoma in situ - heavy vitamin deficiency
* Pregnancy
* less than 18
* Satisfying women
* No tobacco abuse
* satisfying therapy with local immunmodulators in lichen ruber
* surgical therapy of leukoplakia indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Changes in percent (%) of the initial area in mm2 assessed on recall appointment and by a blinded examiner on photographs with a caliper. | each treatment average once a week, recall after 4 weeks

SECONDARY OUTCOMES:
pain due to treatment, assessed by visual analogue scale (VAS) | each treatment, average once a week

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Dvorak, PD, DMD, MD, Study Director — Medical University Vienna
Locations (1):
- Bernhard Gottlieb University Clinic of Dentistry, Vienna, Austria